CLINICAL TRIAL: NCT06351462
Title: Comparative Health Status and Quality of Life of Patients With Sickle Cell Disease (SCD) Who Underwent Matched-sibling Hematopoietic Stem Cell Transplantation Versus Non Transplanted SCD Case-control Patients
Acronym: TRANSPLANTORN2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200008
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Sickle Cell Disease
Keywords: Hematopoietic stem cell transplantation
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients transplanted from allogeneic HLA-compatible sibling donor or from sibling cord blood unit (Other)
  Interventions: Other: Spermogram; Other: Hospital Anxiety and Depression Scale (HADS); Other: SF36 Quality of life questionnaire; Other: Psychologist interview; Other: Optional sera banking; Other: Optional DNA banking
- Controlled patients - not transplanted (Other)
  Interventions: Other: Spermogram; Other: Hospital Anxiety and Depression Scale (HADS); Other: SF36 Quality of life questionnaire; Other: Psychologist interview; Other: Optional sera banking; Other: Optional DNA banking

INTERVENTIONS:
Other: Spermogram — Spermogram will be proposed to men
Other: Hospital Anxiety and Depression Scale (HADS) — Anxiety and depression will be evaluated 10 years after HSCT
Other: SF36 Quality of life questionnaire — Quality of life will be evaluated 10 years after HSCT
Other: Psychologist interview — During a follow-up visit
Other: Optional sera banking — One in the study
Other: Optional DNA banking — Once in the study

SUMMARY:
The long term burden of morbidity and mortality in the natural history of sickle cell disease has not been compared up to date to the risks and mortality of a curative option like bone marrow transplantation in severe sickle-cell disease patients. Given this lack of data, primary-care Sickle Cell Disease (SCD) physicians and transplant physicians are prevented from a factual debate over the benefit/risk ratio for each patient and refining indications of transplant in patients. Therefore, the present study seeks to describe and compare the very long-term outcomes after either Human Leukocyte Antigen (HLA) -matched sibling transplantation (study arm) and "non-transplant care" for severe sickle cell disease SCA patients in order to yield robust comparative data regarding both arms.

The main objective is to assess the benefit of Hematopoietic stem cell transplantation (HSCT) regarding quality of life compared to standard care after 10 years, in patients with severe Sickle Cell Disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

Study population (exposed-patients), all criteria should be fulfilled:

1. Patients alive with Sickle Cell Anemia (SCA, meaning SS and Sbeta0 sickle cell anemia genotype)
2. Patients transplanted from allogeneic HLA-compatible sibling donor or from sibling cord blood unit from the 1st of January 2000 and the 31st of December 2012, whatever the age at transplant
3. Patients having received conditioning regimen containing busulfan 1mg/kg/dose (or equivalent adjusted body-weight dosage according to recommendation) x 16 doses + cyclophosphamide 200mg/kg total dose + anti-thymoglobuline
4. For patient under 18 years at time of enrolment, signed informed consent from both parental representatives
5. For patient aged 18 years old : signed informed consent
6. Having an affiliation to a social security regime

Control-population (Non-exposed patients) :

For each allografted patient, one non-exposed patient will be matched, based on the following criteria:

* Gender
* Age at the date of transplantation of the exposed patient (+/- 1 year)
* Foetal hemoglobin (HbF) level (+/- 3%) before treatment intensification (defined as the initiation of either hydroxyurea or a transfusion program)
* Hb level (+/- 0,9 g/dl) before treatment intensification

  1. For patient under 18 years at time of enrolment, signed informed consent from both parental representatives
  2. For patient above 18 years of age: signed informed consent
  3. Having an affiliation of to a social security regime

Exclusion Criteria:

Study population:

* Transplantation from donor other than sibling or related cord-blood
* Conditioning regimen other than busulfan 16mg/kg total dose + cyclophosphamide 200mg/kg total dose + anti-thymoglobuline

For both population:

* Absence of signed informed consent
* Having any debilitating medical or psychiatric illness, which preclude understanding of the inform consent as well as optimal treatment and follow-up

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life assessed by SF36 | 10 years after HSCT
  It will be assessed by the Short-form 36 (SF36) scale. The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The Medical Outcomes Study 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.

SECONDARY OUTCOMES:
Evaluation of gonadal function | 10 years after HSCT
  Spermogram in men (proposed not requested), Luteinising Hormone (LH), Follicle-Stimulating Hormone (FSH), estrogen, Anti-Müllerian Hormone (AMH) in women, testosterone in men, Amenorrhea in women.
Evaluation of quality of life | 10 years after HSCT
  Questionnaire including data about employment, education level, social financial support.
Proportion of patients with anxiety and depression | 10 years after HSCT
  Anxiety and depression levels will be assessed using the Hamilton Anxiety Depression scale : The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11)

IPD SHARING:
Plan to Share IPD: Undecided